CLINICAL TRIAL: NCT01767818
Title: Longitudinal, Single-center Prospective Study to Assess Progression of Clinical Features and Biologic Markers of Parkinson's Disease Subjects of Varying Levels of Disease Severity
Brief Title: Parkinson's Disease Biomarker Program
Acronym: PDBP
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: NS-12-011; 1U01NS082148-01 (NIH)
Record Dates: First submitted 2013-01-07; First posted 2013-01-14 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimen collection from all enrolled patients and cerebrospinal fluid (CSF) from patients who have provided additional and optional consent to CSF collection.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Previously treated PD patients: 220 subjects with PD treated and responsive to dopaminergic medication
- Previously untreated PD: 20 subjects with de-novo, previously untreated PD confirmed by I-123 Ioflupane SPECT
- Healthy age-matched controls: 46 age-matched healthy controls will be studied.

SUMMARY:
The primary objective of this study is to obtain detailed clinical information and biologic specimens from subjects with PD toward the ultimate end of identifying a biomarker of PD. Because of the inherent difficulties of using clinical outcome measures to assess disease modification, the identification of biomarkers of PD is of paramount importance. The ideal PD biomarker would be one that is easily assayed in a convenient biological sample, varies proportionally with disease severity, is abnormal during the pre-symptomatic phase of the illness, and is unaffected by drugs or other interventions used to treat PD. The existence of a sensitive biomarker with these properties would enable much more effective disease modifying research that would likely be able to take advantage of smaller and potentially shorter trials.

DETAILED DESCRIPTION:
Subjects will be asked to attend study visits every 6 months for up to 5 years of follow up. Each visit will consist of patient outcomes questionnaires, neurological exams, computerized assessments of gait and balance, a video recorded motor exam, and biological specimen collection for biomarker discovery.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic PD meeting UK PD Society Brain Bank Criteria (Step 1, Step 2, and 2 items present from step 3).1
* Male or female age 30 years or older at time of PD diagnosis, Hoehn & Yahr (H&Y) stage I-IV.
* Confirmation from I-123 Ioflupane SPECT (DatScan®) of dopamine transporter deficit for de-novo, untreated patients.
* Clinical evidence of response to dopaminergic medication (MAO-B inhibitors, dopamine agonists, levodopa, or combinations) in patients on treatment for PD.
* Ability to provide written informed consent in accordance with Good Clinical Practice (GCP), International Conference on Harmonization (ICH), and local regulations.
* Able to make visits to UT Southwestern every 6 months for up to 5 years without undue hardship.

Exclusion Criteria:

* Idiopathic PD, H&Y stage 5, as these will be unable to participate in gait assessments.
* Confirmed or suspected atypical parkinsonian syndromes due to drugs, metabolic disorders, encephalitis, or degenerative diseases.
* Presence of definite dementia (MoCA < 17)2.
* For de-novo subjects: received any of the following drugs that might interfere with dopamine transporter SPECT imaging: neuroleptics, metoclopramide, alpha methyldopa, methylphenidate, reserpine, or amphetamine derivative, within 6 months of screening.
* For the prospective CSF cohort: current treatment with anticoagulants (e.g., coumadin, heparin) that might preclude safe completion of the lumbar puncture.
* For the prospective CSF cohort: any condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or known clinically significant coagulopathy or thrombocytopenia.
* Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (1) de-novo, previously untreated patients within 5 years of symptom onset, n=20, and (2) patients on treatment with and clinically responsive to MAO-B inhibitors, dopamine agonists, amantadine, or levodopa (or combinations), n=220 and (3) healthy control patients without evidence of degenerative nerological disease.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2012-11; Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
To estimate the mean rates of change and the variability around the mean of clinical outcomes in PD patients over 3-5 years of follow-up comparing these rates between PD patients of each stage of the Hoehn and Yahr. | 5 years
  This analysis will evaluate rates of progression in PD subjects and determine predictors of fast vs. slow progression

SECONDARY OUTCOMES:
To determine the predictive value of iTUG/iSWAY test results on future course of the disease | 5 years
  This analysis aims to determine if automated gait or balance parameters can classify PD subjects as fast vs slow progressors, and whether gait or balance parameters can track disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dewey, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Sethi A, Dilwali S, McCreary M, Dewey RB Jr. Oral Levodopa Formulation Does Not Affect Progression of Parkinson Disease. Clin Neuropharmacol. 2021 Mar-Apr 01;44(2):47-52. doi: 10.1097/WNF.0000000000000437. PMID 33538517
- See also: Parkinson's Disease Biomarker Program Official Website — http://pdbp.ninds.nih.gov/